CLINICAL TRIAL: NCT02476149
Title: Biomechanical Properties of Keratoconic Eyes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Dr Phillip J Buckhurst, Associate Professor, University of Plymouth
Other Study IDs: 15/SW/0107
Record Dates: First submitted 2015-06-14; First posted 2015-06-19 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Corneal Cross-linking — All participants recruited for the study will be scheduled for corneal crosslinking treatment

SUMMARY:
In keratoconus (KC) corneal thinning and protrusion can cause myopia and irregular astigmatism, affecting vision. The biomechanical properties of the cornea is maintained by an intricate collagen network, which is responsible for its shape and function. In KC this collagen network is disrupted resulting in the cornea losing its shape and function. Keratoconic changes are focal and localised to certain regions of the cornea and the early detection of these changes is challenging. Screening methods include corneal topography (evaluation of anterior corneal surface curvature), tomography (assessing the morphological features of the anterior segment) and aberrometry (measuring the optical aberrations of the eye). More recent research suggests that the biomechanical destabilization of the cornea may precede topographic and tomographic evidence of KC. Management of KC depends on disease severity with severe cases being treated with keratoplasty and less severe cases with cornealcollagencrosslinking (CXL). CXL is an emerging technique, which aims to increase the biomechanical strength of the keratoconic cornea. Despite strong evidence of changes in the biomechanical properties in human corneas following CXL, there is a significant need for accurate measures of biomechanical changes in vivo pre and post CXL. Until recently technical limitations have restricted the ability to assess the biomechanical properties of the whole cornea in vivo. With the introduction of the CorvisST (Oculus) it is now possible to assess regional biomechanical behaviour of the cornea. The output from the device provides a variety of parameters to indicate the cornea's biomechanical strength. To date, the association between the deflection behaviours in various regions of the cornea in keratoconic eyes preand post CXL has not been studied. In order to effectively assess the clinical benefits of CXL such information is vital. The primary goal of this investigation is to investigate regional biomechanical properties of the keratoconic eye before and after CXL.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects over the age of 18 with keratoconus who are enrolled for collagen crosslinking treatment

Exclusion Criteria:

* Any patient who has had surgical complications will also be excluded from participation in the study.

Determination during enrolment:

* Pregnancy or breastfeeding during the study
* Any kind of systemic disease which affect collagen and the body water regulation system (Marfan syndrome, osteogenesis imperfect, pseudozanthoma elasticum, EhlersDanlos, diabetes, rosacea, acne, cardiovascular disease, thyroid disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified as those patients who are due to undergo corneal collagen crosslinking treatment
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change of the corneal hysteresis following corneal crosslinking (mmHg) | Up to 3 months prior to corneal collagen crosslinking treatment and at 3-6 months after treatment
  Corneal hysteresis as measured using the CorvisST

SECONDARY OUTCOMES:
Change of refractive error following corneal crosslinking (LogMAR) | Up to 3 months prior to corneal collagen crosslinking treatment and at 3-6 months after treatment
  Refractive error measured using objective refraction
Axial Length prior to corneal crosslinking (mm) | Up to 3 months prior to corneal collagen crosslinking treatment
  Axial length determined with the LenStar
Axial Length axial length following corneal crosslinking (mm) | At 3-6 months after treatment
  Axial length determined with the LenStar
Change in corneal curvature following corneal crosslinking (mm) | Up to 3 months prior to corneal collagen crosslinking treatment and at 3-6 months after treatment
  Corneal curvature assessed with the Pentacam HR
Tear break up time prior to corneal crosslinking (s) | Up to 3 months prior to corneal collagen crosslinking treatment
  Tear break up time determined using the Oculus K5
Tear break up time following corneal crosslinking (s) | At 3-6 months after treatment
  Tear break up time determined using the Oculus K5

CONTACTS AND LOCATIONS:
Locations (1):
- Plymouth University, Plymouth, Devon, United Kingdom